CLINICAL TRIAL: NCT04019587
Title: Cross-Cultural Adaptation and Psychometric Properties of the Fear of Falling Avoidance Behaviour in Turkish Community-dwelling Older Adults
Brief Title: Turkish Version of Fear of Falling Avoidance Behavior Questionnaire
Status: Completed | Type: Observational
Sponsor: Ordu University (Other)
Responsible Party: Principal Investigator, Sevim ACARÖZ CANDAN, Head of Department of Physiotherapy and Rehabilitation, Ordu University
Other Study IDs: OrduU5
Record Dates: First submitted 2019-07-11; First posted 2019-07-15 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2019-12

CONDITIONS: Fall; Fear; Older People

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Test of reliability and validity
  Interventions: Diagnostic Test: Fear of Falling Avoidance Behavior Questionnaire administration

INTERVENTIONS:
Diagnostic Test: Fear of Falling Avoidance Behavior Questionnaire administration — The Questionnaire includes 14 items dealing with avoidance behavior. All items will be asked by face to face technique.

SUMMARY:
This study is planned to translate the Fear of Falling Avoidance Behaviour Questionnaire (FFABQ) into Turkish and to assess the psychometric properties (validity, reliability, responsiveness, floor and ceiling effect) of this Turkish version.

DETAILED DESCRIPTION:
The permission for the Turkish version was received by Landers. The translation will be made according to Beaton et al. guidelines. The internal reliability of the FFABQ Türkish version will be assessed using Cronbach's alpha, and item analyses will be conducted by examining the effect on Cronbach's alpha of excluding each of the six FOG-Q items individually. The test-retest reliability will be assessed using intraclass correlation coefficient (ICC).

Convergent validity will be evaluated by means of Spearman rank correlation coefficient (rs). In this section will be determined the correlation between the Activities-specific Balance Confidence Scale and visual analog scale for fear of falling.

ELIGIBILITY:
Inclusion Criteria:

* having good cognitive functions (Standardized Mini Mental Test score of 24 and above)
* To be able to live independently in the community,
* to voluntarily participate

Exclusion Criteria:

* The use of drugs that may affect balance
* Polypharmacy status
* Having serious musculoskeletal or neurological disorders,
* Lower or upper limb amputation that may affect balance.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Community dwelling older adults
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2019-07-15 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Fear of Falling Avoidance Behavior Questionnaire (FFABQ) | 7 minutes
  The FFABQ quantifies avoidance behavior (activity limitation and participation restriction) related to the fear of falling. It consists of 14 items ranked using the Likert-style, 5-point ordinal scale as described above, resulting in a total possible score of 56 points. A high score indicates greater activity limitation and participation restriction as a result of the fear of the falling.

SECONDARY OUTCOMES:
Activities-specific Balance Confidence (ABC) | 10 minutes
  The Activity-specific Balance Confidence (ABC) Scale is commonly recommended for evaluating the person's confidence related to fear of falling.The ABC scale contains 16 items to assess balance confidence in performing simple to complex activities, such as walking around the house, stepping onto an escalator, and walking outside on an icy sidewalk.6,22 The total score of ABC scale ranges from 0% - 100%, where 0% means "not confident" and 100% means "completely confident".22 The confidence scores could be interpreted in a categorical fashion of high (> 80%), moderate (50 - 80%) and low (< 50%) levels of physical functioning.
Visual Analog Scale (VAS) for Fear of Balance | 2 minutes
  10 points VAS will be used to assess the fear of falling. The older adult scores their fear with the number that best expresses the fear of falling. 0 indicates no fear and 10 indicates extreme fear.

CONTACTS AND LOCATIONS:
Overall Officials: Sevim A CANDAN, PhD, Principal Investigator — Ordu University
Locations (1):
- Sevim ACARÖZ CANDAN, Ordu, Altinordu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No